CLINICAL TRIAL: NCT06354452
Title: Preadmission Use of Statin Therapy and Sepsis-related Mortality in ICU Patients: a Population-based Cohort Study.
Brief Title: Effect of Statin Therapy on Sepsis-related Mortality in Intensive Care Unit Patients
Acronym: HGG_UCI1
Status: Completed | Type: Observational
Sponsor: Hospital de Granollers (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Principal Investigator, Josep Maria Badia, Prof, Hospital de Granollers
Other Study IDs: HGG2024_01
Record Dates: First submitted 2024-01-22; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Mortality; Statins; Corticoid
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Association

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a diagnosis of sepsis: All patients with a diagnosis of sepsis admitted to the hospitals of the public hospital network of Catalonia, Spain, were included.
  Interventions: Other: Person-level linkage of the database looking for relationship with sepsis survival and previous intake of certain drug families and previous dependence on health services.

INTERVENTIONS:
Other: Person-level linkage of the database looking for relationship with sepsis survival and previous intake of certain drug families and previous dependence on health services. — A descriptive analysis of the baseline demographics, risk factors, health status, comorbidities, frailty, and previous dependence on health services of all patients admitted to hospitals in the region will be carried out.
  Both the overall data of patients admitted to hospitals in any ward and those admitted to ICU will be analysed. The survival data of patients will be compared with their previous individual drug consumption, trying to find out the relationship between chronic consumption of certain families of drugs and inhospital survival to sepsis. In addition, drug dependence and dependence on health services of sepsis survivors will be studied in comparison with their situation prior to sepsis.

SUMMARY:
The average age of patients with sepsis has increased in recent years in parallel with the incidence of sepsis. Many of these patients are frail and require various medications for the treatment of their chronic diseases. Common treatments, including e.g. sarcopenic drugs (statins, sulphonylureas, methyglinides), antioxidants that prevent sarcopenia (allopurinol) or immunoregulators (corticosteroids) may influence the survival and functional prognosis of these patients. Knowing which drugs influence sepsis survival and to what degree patients who survive sepsis have functional deterioration and increased comorbidity and which modifiable factors limit this may be essential.

DETAILED DESCRIPTION:
The hypothesis of the study is that poor baseline health status, defined by frailty, comorbidities and chronic drug use, determines sepsis survival and long-term functional status of surviving patients. In addition, the study aims to analize the relationship between different groups of drugs, especially sarcopenal drugs, and sepsis survival in patients admitted to hospitals and Intensive Care Units in a region of 8 million inhabitants. Preliminary data suggest that patients with prior corticosteroid use have poorer survival to sepsis, while chronic statin use may be a protective factor.

This will be a retrospective population-based observational analysis of a large cohort of patients with sepsis using a population-based database over a 2-year period.

The data will be obtained from the Catalan Health System (CatSalut) Minimum Basic Data Set (CMBD) registers (compulsory admissions register for all public and private acute care hospitals in Catalonia, Spain. The registry is intended for the evaluation and optimisation of the use of resources, provides support and improves healthcare planning and facilitates the management of purchases and payments. A cohort of approximately 25,000 patients per year is available from the aforementioned databases (2). Data from 2018 and 2019 (pre-pandemic) will be initially included.

Sepsis will be defined using the methodology described by Angus et al, which is currently referenced for population-based studies, consisting of coding a diagnosis of infection with acute organ failure, or sepsis or septic shock.Patients requiring Intensive Care Unit (ICU) admission were identified from the coded procedures of mechanical ventilation, continuous renal replacement techniques (CRRT), tracheostomy, or extracorporeal membrane oxygenation (ECMO).

To analyse outpatient prescriptions, a patient will be considered to have prior treatment with a given medication if, during the 8 months prior to admission for sepsis, a minimum of 6 containers of that drug had been dispensed. The Anatomical, Therapeutic, Chemical (ATC) drug classification of the World Health Organization (WHO) will be used.

An analysis of demographics, risk factors, baseline status, comorbidities, and previous dependence on health services of all patients admitted to hospitals in the region will be carried out. Overall patients admitted to hospitals and those admitted to ICU will be analysed separately. Survival data will be compared with previous drug use, trying to find out the relationship between dependence to some groups of these drugs and survival to sepsis. In addition, drug dependence and health services dependence of sepsis survivors will be studied in comparison with their pre-sepsis situation.

A descriptive analysis of the baseline characteristics of the sample will be performed using absolute values and percentages or mean and standard deviation, as appropriate. To establish the relationship between the dependent and independent variables, a bivariate analysis will be performed using the chi-square or t-Student test, as appropriate. A logistic regression model will be applied to determine the risk factors for mortality, analysing the scores for comorbidities, frailty (defined as emergency admissions, being a resident or institutionalised, being previously defined as a complex chronic patient or advanced chronic disease) and chronic consumption of certain families of drugs, for all those variables that had obtained statistical significance in the bivariate analysis. Statistical significance will be established with a p-value of less than 0.001.

The creation of the scale predictive of mortality will be based on the combination of the risk factors detected in the previous logistic regression analyses. The reliability and validity of the scale for subgroups of the sample will be analysed to check that the psychometric characteristics of the instrument were valid for the different types of population. To study sepsis mortality, Cox regression models or competing risk models will be performed, comparing baseline states and different pharmacological treatments.

The impact on health care consumption of patients who do not survive sepsis will be based on data from the Catalan Health System (CatSalut) Minimum Basic Data Set (CMBD) registers, and it will not be an economic study using cost-effectiveness or health-assessment methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of sepsis admitted to the hospitals of the public hospital network of Catalonia, Spain. Sepsis will be defined using the methodology described by Angus et al., which is currently referenced for population-based studies, consisting of coding a diagnosis of infection with acute organ failure, or sepsis or septic shock.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of sepsis admitted to the hospitals of the public hospital network of Catalonia, Spain, will be included. The data will be obtained from the Catalan Health System (CatSalut) Minimum Basic Data Set (CMBD) registers (compulsory admissions register for all public and private acute care hospitals in Catalonia, Spain, over a 2-year period (2018 and 2019).
Sampling Method: Non-Probability Sample
Enrollment: 59578 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Death due to sepsis | From date of hospital admission until the date of hospital discharge, assessed up to 12 months
  Inhospital death after an episode of sepsis requiring hospital or ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Badia, MD, PhD, Study Director — Hospital General de Granollers
Locations (1):
- Hospital General de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Restrictions apply to the availability of these data, which belong to a national database and is not publicly available.

REFERENCES:
- [Derived] Iglesias R, Badia JM, Vela E, Yebenes JC. Baseline morbidity and chronic medications as determinants of sepsis outcomes: focus on statins, corticosteroids, and NSAIDs in a population-based cohort of 59,578 patients. Front Pharmacol. 2026 Jan 15;16:1727662. doi: 10.3389/fphar.2025.1727662. eCollection 2025. PMID 41625328
- [Derived] Iglesias R, Badia JM, Vela E, Monterde D, Carlos Yebenes J. Influence of comorbidities and chronic medications on ICU mortality in sepsis: A population-based cohort study of 12,095 patients. Med Clin (Barc). 2026 Jan;166(1):107265. doi: 10.1016/j.medcli.2025.107265. Epub 2026 Jan 7. English, Spanish. PMID 41505944